CLINICAL TRIAL: NCT05934656
Title: Gut Research Advancing a Mechanistic and Personalised Understanding of Symptoms in Cystic Fibrosis: The GRAMPUS-CF Strategic Research Centre
Brief Title: Understanding Gut Symptoms in People With Cystic Fibrosis
Acronym: GRAMPUS-CF SRC
Status: Recruiting | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: Cystic Fibrosis Trust (Other); Motilent (Unknown); Nottingham Trent University (Other); Vanderbilt University Medical Center (Other); University of Leeds (Other); Brandenburg Medical School Theodor Fontane (Other); University of Glasgow (Other); National Institute for Health Research, United Kingdom (Other Government); University of Birmingham (Other); Northumbria University (Other); Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: SRC 023
Record Dates: First submitted 2023-05-30; First posted 2023-07-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Cystic Fibrosis; Gastrointestinal Dysfunction
Keywords: Gastrointestinal symptoms; Gastrointestinal transit; Gastrointestinal microbiome; Inflammation; Magnetic Resonance Imaging; Oro-caecal transit time; Small bowel water; Colonic volume; Stool microbiome; Diet; Phenotypes; Biomarkers; Diet quality; Dietary indices; Bloating; Constipation; Malabsorption; Latent class analysis
MeSH Terms: conditions — Cystic Fibrosis; Inflammation; Constipation; Malabsorption Syndromes | interventions — Latent Class Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool samples frozen pre-analysis
  Whole blood samples for the analysis of peripheral blood mononuclear cells (PBMC).
  PBMCs will be stored at -80oC.
  Serum samples stored at -80oC.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People with cystic fibrosis: People with confirmed diagnosis aged over six year old
  Interventions: Other: Latent class analysis

INTERVENTIONS:
Other: Latent class analysis — The investigators will conduct a longitudinal study comprising nested groups A to C of the study population, with progressively more detailed mechanistic investigations. No control group.
  Group A will complete a CF-specific measure of gut symptoms (CFAbd-Score), a generic constipation score (PAC-SYM) and 24 hour dietary recall (Intake24).
  Group B will have stool and blood for microbiome, inflammatory mediators and faecal fat.
  Group C will have gut MRI and exploratory studies of inflammation.

SUMMARY:
Although chest infections affect wellbeing and survival in cystic fibrosis (CF), most people with CF also have difficulty digesting food and must take medication for this. In spite of this treatment, two thirds of people with CF miss school or work because of tummy symptoms (pain, bloating and wind). In some cases these symptoms become severe leading to bowel obstruction and hospital admission. Long term, people with CF have a greater risk of bowel cancer. The investigators asked people with CF and health professionals to suggest the most important questions for research. Treatment of gut symptoms was in their top 10 list. Current treatments are often ineffective because the investigators do not fully understand why symptoms occur. GRAMPUS-CF SRC will describe accurately the categories of gut symptoms in CF and find out why they occur. The investigators will do this using magnetic resonance imaging (MRI) scans and tests which give a detailed description of the germs in the bowel or which measure inflammation. The investigators will also study the effects of diet, using a questionnaire. The investigators will link these results together, using advanced statistics to find the factors causing gut symptoms. The investigators will then identify treatments which are likely to be helpful. In future work the investigators will test these in clinical trials.

DETAILED DESCRIPTION:
This is a multicentre longitudinal observational study Study.

Hypothesis 1 - Distinct phenotypes of gut symptoms in CF can be defined, using symptom questionnaires.

Hypothesis 2 - These phenotypes will be characterised by differences in mechanism, elucidated by MRI physiology, gut microbiome, inflammatory markers and dietary factors.

Hypothesis 3 - Integration of mechanistic data will identify pathways which can be targeted by new and repurposed therapeutics, dietary modifications and biomarkers to identify those patients likely to benefit.

Study Design Tiered study (3 groups), using latent class analysis to characterise phenotypes of CF gut symptoms, from clinical and questionnaire data.

No control group. The investigators will conduct a longitudinal study comprising nested groups A to C of the study population, with progressively more detailed mechanistic investigations.

Group A will complete a CF-specific measure of gut symptoms (CFAbd-Score) and a generic constipation scoring using the 'Patient Assessment of Constipation-Symptoms' (PAC-SYM) and a dietary questionnaire (Intake24). Participants will provide questionnaire data at 3 time points, 6 months apart (baseline, 6 and 12 months).

Group B will have stool and blood for microbiome, inflammatory mediators and faecal fat. Participants will provide stool and blood samples at 3 time points, 6 months apart (baseline, 6 and 12 months).

Group C will have gut MRI and exploratory studies of inflammation (immune gene expression and micro RNA analysis). Participants will spend approximately 6 hours in the MRI scanning suite on a single day.

Group A - 300 adults & 50 children. Group B - 100 adults & 20 children (group B participants will be drawn from group A).

Group C - 40 adults & 10 children (group C participants will be drawn from group B).

Total final enrolment 300 adults & 50 children

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of cystic fibrosis (clinical features of CF combined with either a genotype known to be associated with CF or a diagnostic sweat chloride).
2. For participants enrolled in group A via the mobile phone app, self-reported diagnosis will be accepted.
3. Adult patients will be aged 16 years and over and attend the Nottingham or Leeds CF Centres.
4. Paediatric patients will be aged 6-15 years and attend the Nottingham CF Centre.
5. Capacity to consent, or to understand the requirements of the study where parent or guardian consent is needed.
6. English-speaking (the panel of questionnaires the investigators will use has so far been validated only in English).

Exclusion Criteria:

EXCLUSIONS TO PARTICIPATION IN ANY PART OF THE STUDY

1. Self-reported diagnosis of an additional gastrointestinal condition e.g. inflammatory bowel disease, coeliac disease or gastrointestinal cancer.
2. Patients from Leeds previously enrolled in the IGLOO-CF Study* * Data from the IGLOO-CF Study will form the validation dataset for the latent class analysis in GRAMPUS-CF.

EXCLUSIONS TO PARTICIPATION IN GROUP C (MRI SCANS)

1. Measurement of Forced Expiratory Volume in 1 second (FEV1) of <40% predicted using Global Lung Initiative criteria, according to clinical records.
2. Contra-indication to MRI scanning, such as embedded metal, pacemaker.
3. Unable to stop medications directly prescribed to alter bowel habit, such as laxatives of anti-diarrhoeals, on the study day.
4. Previous resection of any part of the gastro-intestinal tract apart from appendicectomy or cholecystectomy. Surgical relief of distal intestinal obstruction syndrome or neonatal ileus will be permitted unless clinical records show excision of intestine >20cm in length.
5. Intestinal stoma
6. Diagnosis of inflammatory bowel disease or coeliac disease confirmed by biopsy
7. Gastrointestinal malignancy
8. Unable to comply with dietary restrictions required for the study
9. Pregnancy - tests are available at the Sir Peter Mansfield Imaging Centre if participants are unsure.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children aged 6-15 years old and adults aged over 16 years old with cystic fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Identification of distinct phenotypes of gastrointestinal symptoms in people with cystic fibrosis | Baseline
  Latent class analysis will be used to determine symptom clusters (phenotypes). This will depend on the scores on the CF-Abd and Patient Assessment of Constipation symptom (PAC-SYM) questionnaires.
  CF-Abd includes 28 items rated on a 6-poin. The scoring scale is between 0 and 100 with higher values for increasing frequency and/or severity of symptoms.
  PAC-SYM includes 12 items rated on a 5-point (0-4) Likert scale. The global score is the mean of all 12 items. Higher score indicates worse symptoms.
  These, together with the data from the dietary questionnaire (Intake24) will be used in the latent class analysis to determine symptom clusters

SECONDARY OUTCOMES:
Association of clusters (primary outcome) with stool inflammatory markers | through study completion (measured at baseline, 6 and 12 months)
  Association of clusters (primary outcome) with stool inflammatory markers to explore possible mechanisms: Faecal calprotectin and faecal cytokines
Association of clusters (primary outcome) with stool elastase | through study completion (measured at baseline, 6 and 12 months)
  Association of clusters (primary outcome) with stool elastase (a marker of pancreatic exocrine function) to explore possible mechanisms
Association of clusters (primary outcome) with stool fat | through study completion (measured at baseline, 6 and 12 months)
  Association of clusters (primary outcome) with stool fat to explore possible mechanisms.
Association of clusters (primary outcome) with faecal microbiome | through study completion (measured at baseline, 6 and 12 months)
  Association of clusters (primary outcome) with faecal microbiome to explore possible mechanisms.
Association of clusters (primary outcome) with faecal metabolome | through study completion (measured at baseline, 6 and 12 months)
  Association of clusters (primary outcome) with faecal metabolome to explore possible mechanisms
Association of clusters (primary outcome) with blood markers of gut permeability | through study completion (measured at baseline, 6 and 12 months)
  Association of clusters (primary outcome) with blood markers of gut permeability to explore possible mechanisms.
Association of clusters (primary outcome) with Magnetic Resonance Imaging metrics | During procedure
  Association of clusters (primary outcome) with Magnetic Resonance Imaging metrics to explore possible mechanisms: small bowel water content, orocaecal transit time, colonic volume and motility

CONTACTS AND LOCATIONS:
Overall Officials: Alan Smyth, Principal Investigator — University of Nottingham
Locations (1):
- Nottingham University Hospitals Trust, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Applications will be considered for access to study data, with no participant identifiers.
Time Frame: Applications will be considered from the time that our own data analysis is complete (expected to be 31/12/26), for a maximum of 7 years after study completion.
Access Criteria: Requests should be addressed to the chief investigator via the study email address (grampuscf@nottingham.ac.uk). Requests will be assessed on a case-by-case basis.
  Applications should state the research question being addressed and include a link to the researcher's published protocol. This will be reviewed by the research team and a final decision to share data will be the responsibility of the chief investigator. Data sharing is specifically mentioned in the participant information sheet and consent for this has been obtained.

REFERENCES:
- See also: The Cystic Fibrosis Trust Strategic Research Centres — https://www.cysticfibrosis.org.uk/the-work-we-do/research/gut-research-advancing-a-mechanistic-and-personalised-understanding-of